CLINICAL TRIAL: NCT05658055
Title: The Effect of Probiotics With Vonoprazan-amoxicillin Dual Therapy on Gut Microbiotain After Helicobacter Pylori Eradication: A Randomized Controlled Trial
Brief Title: The Effect of Probiotics on Gut Microbiotain After Helicobacter Pylori Eradication
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Director of Gastroenterology, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20221124-08
Record Dates: First submitted 2022-12-06; First posted 2022-12-20 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Helicobacter Pylori Infection; Infections; Intestinal Bacteria Flora Disturbance
MeSH Terms: conditions — Infections | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin combined with vonoprazan (Active Comparator): The subjects will be given 20mg vonoprazan twice a day and 1000mg amoxicillin three times a day. These two drugs were taken continuously for 14 days
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin
- Probiotics combined with vonoprazan and amoxicillin (Experimental): The subjects will be given 20mg vonoprazan twice a day, 1000mg amoxicillin three times a day and probiotics three times a day. These three drugs were taken continuously for 14 days.
  Interventions: Drug: Vonoprazan; Drug: Amoxicillin; Drug: probiotics

INTERVENTIONS:
Drug: Vonoprazan — Potassium-competitive acid blocker
Drug: Amoxicillin — Antibiotic for H. pylori eradication
Drug: probiotics — Medilac-S; Enterococcus faecium 4.5*10^8 and Bacillus subtilis 5.0*10^7, Hanmi,Beijing, China
  Arms: Probiotics combined with vonoprazan and amoxicillin

SUMMARY:
The purpose of this study is to evaluate the effect of probiotics during vonoprazan-amoxicillin dual therapy on the gut microbiota in Helicobacter pylori eradication and to investigate whether the eradication rate of H.pylori will be improved when adding probiotics

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will undergo a 1-week screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirement will be included in this simultaneous blind test. A total of 100 patients with HP infection were enrolled in this study. All patients were randomly divided into two groups according to the ratio of 1:1. Group A was given vonoprazan 20mg bid, amoxicillin 1000mg tid, Probiotics 3tabltes tid for 14 consecutive days; Group B was given vonoprazan 20mg bid and amoxicillin 1000mg tid for 14 days. On the 14th days of treatment, the researchers will follow up the patients' adverse reactions and medication compliance. The feces of the subjects were collected one day before the treatment, and on the 14th and 42th days after the treatment; After 4 weeks of drug withdrawal, all subjects will be reexamined with 13C-UBT.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18 and 65 years; Sexes eligible for study: both;
2. patients who are diagnosed with Helicobacter pylori;
3. treatment-naive patients or patients who failed to eradicate Helicobacter pylori in the past but haven't undergone eradication therapy in the past six months;
4. voluntary to be involved in the study and written informed consent was obtained from all patients

Exclusion Criteria:

1. allergic reactions to the study drugs;
2. patients with peptic ulcer;
3. patients who underwent eradication therapy for Helicobacter pylori during the last six months;
4. patients who took antibiotics,bismuth agents,probiotics within four weeks prior to treatment and those who took H2 receptor antagonists,proton pump inhibitors(PPIs) or potassium competitive acid blockers within two weeks prior to treatment;
5. patients who are taking glucocorticoids, non-steroidal anti-inflammatory drugs or anticoagulants;
6. patients who have history of esophageal or gastric surgery;
7. pregnant or lactating women;
8. patients who have severe concurrent diseases such as hepatic,cardiovascular,respiratory,renal disorders or malignancies;
9. Alcohol abusers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The comparison of the gut microbiota composition | 12mouth
  Stool samples were collected at the points of before eradication, after eradication and at confirmation. The gut microbiota composition of individuals was analyzed by 16S rRNA gene sequencing. Microbiome bioinformatics were performed with QIIME2 and R packages.

SECONDARY OUTCOMES:
Helicobacter pylori eradication rate | four to six weeks after completion of the medication
  Helicobacter pylori Eradication will be determined by ¹³C-urea breath test four to six weeks after completion of the medication. The eradication rates will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis.
Adverse event | one week after completion of the medication
  adverse events are recorded by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Zhang, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No